CLINICAL TRIAL: NCT04654143
Title: A Phase I, Double-blind, Randomized, Placebo-controlled Study to Investigate the Safety, Tolerability and Pharmacokinetics and Food Effect of BVL-GSK098 Administered as Single and Multiple Oral Doses to Healthy Volunteers
Brief Title: Clinical Trial to Investigate the Safety, Tolerability and Pharmacokinetics of BVL-GSK098 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioVersys AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BVL-GSK098
Record Dates: First submitted 2020-11-15; First posted 2020-12-04 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2022-06

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single Ascending Dose (SAD) (Experimental): There are multiple dose levels or cohorts. Each cohort has 6 subjects randomized to BVL-GSK098 and 2 subjects randomized to placebo.
  Interventions: Drug: BVL-GSK098 capsule, placebo
- Multiple Ascending Dose (MAD) (Experimental): There are multiple dose levels or cohorts. Each cohort has 6 subjects randomized to BVL-GSK098 and 2 subjects randomized to placebo.
  Interventions: Drug: BVL-GSK098 capsule, placebo
- Food Effect (Experimental): This cohort has 6 subjects randomized to BVL-GSK098 and 2 subjects randomized to placebo. Each participant will receive a single oral dose of BVL-GSK098 or placebo administered after the participant eats a high-fat, high calorie breakfast.
  Interventions: Drug: BVL-GSK098 capsule, placebo

INTERVENTIONS:
Drug: BVL-GSK098 capsule, placebo — Oral QD

SUMMARY:
This is a phase I single-center, double-blind, randomized, placebo-controlled study to investigate the safety, tolerability and pharmacokinetics and food effect of BVL-GSK098 administered as single and multiple oral doses to healthy volunteers

DETAILED DESCRIPTION:
This is an exploratory, first-in-human (FIH), double-blind, randomized, placebo-controlled, single and multiple ascending oral dose study in healthy volunteers.The study will be divided into two parts that will be conducted sequentially. Part A is a SAD study to determine the safety, tolerability and PK of single oral doses of BVL-GSK098 in healthy volunteers. In addition, the last cohort of Part A will investigate the effect of food on the PK of BVL-GSK098. Part B is a MAD study to determine the safety, tolerability and PK of BVL-GSK098 following multiple daily oral doses in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteers aged 18 to 55 years inclusive and between 19 and 30 kg/m2 body mass index (BMI) with a minimum weight of 50 kg or men and 45 kg for women, at the time of signing the informed consent.
2. Volunteers who are healthy as determined by the investigator based on medical evaluation including medical history, physical examination and cardiac monitoring.
3. Volunteers who have a clinically acceptable temperature, blood pressure and pulse rate in supine and standing position (systolic blood pressure between 100-140 mm Hg/ diastolic blood pressure between 50-90 mm Hg / HR between 50-100 bpm). Blood pressure and pulse will be measured after a minimum of 3 minutes of resting.
4. Volunteers whose clinical laboratory test results are not clinically relevant and are acceptable to the Investigator.
5. Male volunteers must use appropriate contraception (e.g. condoms as part of a double barrier method) from the time of the first dose until 3 months after the post-study visit.
6. A female volunteer is eligible to participate if she is of non-childbearing potential, defined as:

   1. Is equal to or older than 45 years of age and has not had menses for greater than 1 year,
   2. Amenorrheic for less than 2 years without a hysterectomy and oophorectomy and a follicle-stimulating hormone value in the postmenopausal range upon pretrial (screening) evaluation,
   3. Whose status is post hysterectomy, oophorectomy or tubal ligation.
7. Nonsmokers (i.e., one who has abstained from use of tobaccco and other nicotine-containing products for the last 6 months).
8. Willingness to stay in the investigational site for up to 11 days.
9. Volunteers are capable of giving signed informed consent which included compliance with the requirements and restrictions listed in the consent form and in this protocol.

Exclusion Criteria:

1. Women of childbearing potential
2. Pregnant or lactating women
3. Men with female partners who are lactating or are pregnant
4. Glomerular Filtration Rate (GFR) < 90 mL/min/1.73m2 as calculated by the Chronic Kidney Disease Epidemiology Collaboration formula.
5. Alanine aminotransferase (ALT), Gamma glutamyl transferase (GGT), Aspartate aminotransferase (AST), alkaline phosphatase or serum bilirubin levels must not exceed the upper limit of normal (ULN)
6. A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
7. A positive test for HIV antibody.
8. A positive pre-study drug/alcohol screen.
9. Volunteers who consume more than 21 units of alcohol per week or who have a significant history of alcoholism or drug/chemical abuse (one unit of alcohol equals ½ pint [285 mL] of beer or lager, one glass [125 mL] of wine, or 30 mL of 40% of alcohol by volume distilled spirits).
10. Volunteers who are study site employees, or immediate family members of a study site or sponsor employee.
11. Volunteers with ECG abnormalities (history, or evidence of second-degree heart block of Mobitz type II, third degree heart block, or any abnormality considered relevant by the Investigator), QTcB or QTcF >450 ms or PR>220 ms).
12. Volunteers with a history of additional risk factors for torsade de pointes (TdP) (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)
13. History of clinically significant cardiovascular, renal, hepatic, chronic respiratory or gastrointestinal disease, neurological or psychiatric disorder, as judged by the investigator.
14. History of seizures.
15. Volunteers who have received any prescribed systemic or topical medication within 4 weeks of the first dose administration.
16. Volunteers who have used any non-prescribed systemic or topical medication (including herbal remedies) or megadose vitamins (i.e. 20 to 600 times the recommended daily supplement dose) within 7 days of the first dose administration, unless in the opinion of the Investigator the medication will not interfere with the study procedures or compromise safety.
17. Volunteers who have received any medications, including St John's Wort, known to chronically alter drug absorption or elimination processes within 30 days of the first dose administration.
18. Volunteers who have participated in other clinical trials during the previous 90 days (drug to drug period) in which an investigational drug or a commercially available drug was tested.
19. Exposure to more than 4 new chemical entities in the last 12 months before the first dosing day in this study.
20. Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56-day period.
21. Failure to satisfy the investigator of fitness to participate for any other reason

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2023-01-16 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) and Serious AEs (SAEs) | From screening visit (Day -3 to -30) to end of study (7-10 days post last dose)
  All AEs will be counted and described within each cohort/dose level, by treatment received and tabulated.
Number of participants with clinically significant abnormal findings in hematology parameters | Day 1 until end of study (7-10 days post last dose)
  Blood samples will be collected for the assessment of hematology parameters.
Number of participants with clinically significant abnormal findings in clinical chemistry parameters | Day 1 until end of study (7-10 days post last dose)
  Blood samples will be collected for the assessment of chemistry parameters.
Number of participants with urinalysis findings | Day 1 until end of study (7-10 days post last dose)
  Urine samples will be collected for the assessment of urinalysis parameters.
Number of participants with clinically significant abnormal findings in vital signs | Day 1 until end of study (7-10 days post last dose)
  Number of participants with abnormal vital signs will be assessed.
Number of participants with clinically significant abnormal findings in Electrocardiogram (ECG) Parameters | Day 1 until end of study (7-10 days post last dose)
  Triplicate 12-lead ECGs will be obtained

SECONDARY OUTCOMES:
Maximum observed plasma drug concentration (Cmax) of BVL-GSK098 | Single dose: up to 72 hours; Multiple dose: up to 10 days
  Blood samples will be collected to evaluate Cmax of BVL-GSK098
Time to maximum observed plasma drug concentration (tmax) of BVL-GSK098 | Single dose: up to 72 hours; Multiple dose: up to 10 days
  Blood samples will be collected to evaluate tmax of BVL-GSK098
Area under the plasma drug concentration versus time curve (AUC) of BVL-GSK098 | Single dose: up to 72 hours; Multiple dose: up to 10 days
  Blood samples will be collected to evaluate AUC of BVL-GSK098
Apparent terminal half-life (t1/2) of BVL-GSK098 as appropriate | Single dose: up to 72 hours; Multiple dose: up to 10 days
  Blood samples will be collected to evaluate t1/2 of BVL-GSK098
The effect of food on the plasma concentrations of BVL-GSK098 | up to 72 hours
  Blood samples will be collected to evaluate the food effect on plasma concentrations of BVL-GSK098
Observed accumulation ratio following BVL-GSK098 repeat dosing | up to 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Rosa M Antonijoan, MD, Principal Investigator — Institut de Recerca de l'HSCSP. IIB Sant Pau.
Locations (2):
- Spain (2):
  - CIM Sant Pau, Barcelona
  - Hospital Universitario de La Princesa, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pieren M, Abaigar Gutierrez-Solana A, Antonijoan Arbos RM, Boyle GW, Davila M, Davy M, Gitzinger M, Husband L, Martinez-Martinez MS, Mazarro DO, Pefani E, Penman SL, Remuinan MJ, Vlasakakis G, Zeitlinger M, Dale GE. First-in-human study of alpibectir (BVL-GSK098), a novel potent anti-TB drug. J Antimicrob Chemother. 2024 Jun 3;79(6):1353-1361. doi: 10.1093/jac/dkae107. PMID 38656557